CLINICAL TRIAL: NCT03278717
Title: International Phase III Randomised Study to Evaluate the Efficacy of Maintenance Therapy With Olaparib and Cediranib or Olaparib Alone in Patients With Relapsed Ovarian Cancer Following a Response to Platinum-based Chemotherapy
Brief Title: Study Evaluating the Efficacy of Maintenance Olaparib and Cediranib or Olaparib Alone in Ovarian Cancer Patients
Acronym: ICON9
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL/14/0795
Record Dates: First submitted 2017-07-31; First posted 2017-09-12 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-06

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib; cediranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Olaparib and Cediranib (Experimental): Patients will receive oral olaparib 300mg BD and oral cediranib 20mg OD.
  Patients will attend hospital for a 2 weekly review for the first 8 weeks, then 4 weekly for year 1 and 8 weekly for year 2 onwards until discontinuation of all trial drugs. Treatment may continue beyond progression until the next line of treatment if the patient is deemed to still be deriving clinical benefit. QOL instruments will be collected at baseline, every clinic visit and continue to be completed after relapse.
  Interventions: Drug: Olaparib; Drug: Cediranib
- Olaparib (Active Comparator): Patients will receive oral olaparib 300mg BD.
  Patients will attend hospital for a 2 weekly review for the first 8 weeks, then 4 weekly for year 1 and 8 weekly for year 2 onwards until discontinuation of all trial drugs. Treatment may continue beyond progression until the next line of treatment if the patient is deemed to still be deriving clinical benefit. QOL instruments will be collected at baseline, every clinic visit and continue to be completed after relapse.
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Olaparib is a PARP inhibitor, targeting DNA repair processes.
Drug: Cediranib — Cediranib is an inhibitor of vascular endothelial growth factor-A (VEGF), targeting angiogenesis.
  Arms: Olaparib and Cediranib

SUMMARY:
ICON 9 will assess the efficacy, safety and tolerability of maintenance olaparib in combination with cediranib compared to maintenance olaparib alone following a response to platinum-based chemotherapy in women with relapsed platinum-sensitive ovarian, fallopian tube or peritoneal cancer. Prognostic and predictive factors will be studied from tumour and blood samples.

DETAILED DESCRIPTION:
ICON9 is an international multicentre randomised, phase III trial assessing maintenance treatment with olaparib and cediranib or olaparib alone in women with relapsed ovarian cancer whose disease progressed more than 6 months after first line chemotherapy. Women whose disease responds to platinum chemotherapy following 3 to 4 cycles can be registered for collection of germline BRCA test results if known, and somatic BRCA testing of archival tumour specimens or secondary debulking tissue if required. Patients who have completed treatment and whose disease has responded (partial or complete) to a minimum of 4 cycles of platinum based chemotherapy will be randomised to maintenance treatment of either olaparib and cediranib or olaparib alone.

The maintenance regimen may be continued beyond radiological progression until trial closure if the patient is deemed to still be deriving clinical benefit, but must be discontinued once subsequent treatment is instituted.

ELIGIBILITY:
Registration Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures and the ability to comply with the protocol for the duration of the study, including undergoing treatment and scheduled visits and examinations.
2. Females aged ≥ 18 years with previous histologically proven diagnosis of high grade serous or endometrioid carcinoma of the

   * Ovary
   * Fallopian tube
   * or peritoneum, progressing >6 months after day 1 of the last cycle of first-line platinum-based chemotherapy and requiring treatment with platinum-based chemotherapy on the basis of radiological evidence of disease or following surgical resection of recurrent disease.
3. Patients must have had CT or MRI proven relapsed disease (measureable or non-measureable abnormalities supported by GCIG CA125 criteria of progression), or have had debulking surgery for first relapse.
4. Patients showing evidence of response to chemotherapy mid-treatment (post 3 or 4 cycles), either by CA125 or CT/MRI scan, should be approached for ICON9 trial registration to allow for BRCA mutation status to be assessed (germline and/ or somatic). Patients who underwent surgical debulking must show no evidence of disease progression by the assessments above (CA125 and CT/MRI scan) in order to be approached for registration.
5. Prior front-line maintenance therapy with bevacizumab is permitted.
6. ECOG performance status 0-1.
7. Formalin fixed, paraffin embedded (FFPE) archival/diagnostic tumour sample or from secondary debulking surgery with adequate neoplastic cell content (>30%), must be available for central BRCA testing. For inclusion in i) the genetic HRD Test and ii) the biomarker research, patients must complete the consent form. Translational blood samples are also required, see Laboratory Manual for further details.
8. Patients should have a life expectancy ≥ 16 weeks.
9. Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days prior to study treatment and confirmed prior to treatment on day 1.

   Postmenopausal is defined as age ≥60 years, or:
   * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
   * Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post-menopausal range for women under 50
   * Radiation-induced oophorectomy with last menses >1 year ago
   * Chemotherapy-induced menopause with >1 year interval since last menses
   * Surgical sterilisation (bilateral oophorectomy or hysterectomy)
10. Adequately controlled blood pressure (systolic blood pressure [SBP] ≤140 mmHg; diastolic blood pressure [DBP] ≤ 90mmHg) on maximum of 2 antihypertensive medications.
11. Adequately controlled thyroid function, with no symptoms of thyroid dysfunction.

Randomisation Inclusion Criteria:

1. Patients must have received at least 4 cycles, and a maximum of 6 cycles of second-line platinum-based chemotherapy.
2. In patients with measurable disease, end of treatment scans must have a RECIST v1.1 'partial response' or 'complete response' and meet one of the following CA125 requirements:

   1. If the first screening CA125 value is below the ULN the patient is eligible for randomisation and a second CA125 assessment is not required.
   2. If the first screening CA125 value is greater than ULN then a second assessment is required at least 7 days after the first to confirm eligibility. If the second CA125 value has risen by ≥ 15% then the patient will not be eligible.
3. In patients with non-measurable disease, who have not undergone debulking surgery, they must have had a GCIG CA125 response to chemotherapy and meet one of the following CA125 requirements:

   1. If the first screening CA125 value is below the ULN the patient is eligible for randomisation and a second CA125 assessment is not required.
   2. If the first screening CA125 value is greater than ULN then a second assessment is required at least 7 days after the first to confirm eligibility. If the second CA125 value has risen by ≥ 15% then the patient will not be eligible.
4. Patients who have had debulking surgery at first relapse must have no evidence of disease progression on imaging (CT or MRI) and meet one of the following CA125 requirements:

   1. If the first screening CA125 value is below the ULN the patient is eligible for randomisation and a second CA125 assessment is not required.
   2. If the first screening CA125 value is greater than ULN then a second assessment is required at least 7 days after the first to confirm eligibility. If the second CA125 value has risen by ≥ 15% then the patient will not be eligible.
5. Expected to be able to commence treatment within 7 days post randomisation, and within 4-8 weeks post day 1 of the last cycle of chemotherapy.
6. Adequate bone marrow function as defined below:

   * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/l
   * Platelet (Plt) ≥ 90 x 109/l
   * Haemoglobin (Hb) ≥ 100g/l required and no packed blood transfusions in the 14 days prior to starting trial treatment
7. Adequate liver function as defined below:

   * Serum bilirubin ≤ 1.5 x ULN (or ≤ 3 for cases of known Gilbert's syndrome)
   * Serum transaminases ≤3 x ULN
   * Serum transaminases ≤ 5 x ULN if liver metastasis present
8. Adequate renal function as defined below:

   • Serum creatinine ≤ 1.5 x ULN and calculated glomerular filtration rate (GFR) ≥50ml/min (calculated as per local practice using Wright or Cockroft-gault formula)
9. Urine dipstick for proteinuria <2+. If urine dipstick is ≥ 2+ on two occasions more than one week apart then a 24-hour urine must demonstrate ≤ 1 g of protein in 24 hours or protein/creatinine ratio < 1.5.
10. Adequately controlled blood pressure (systolic blood pressure [SBP] ≤140 mmHg; diastolic blood pressure [DBP] ≤ 90mmHg) on maximum of 2 antihypertensive medications.
11. Germline and/or somatic BRCA mutation status must be known prior to randomisation.

Exclusion Criteria:

1. Non-epithelial ovarian cancer, carcinosarcoma, clear cell carcinoma and mucinous carcinomas.
2. Arterial thrombotic event (including transient ischemic attack, cerebrovascular accident, and peripheral arterial embolus) within the last 12 months.
3. Patients unable to swallow orally administered medication and patients with gastrointestinal impairment that could affect ability to take, or absorption of oral medicines including sub-acute or complete bowel obstruction.
4. Clinically significant signs and/or symptoms of bowel obstruction within 3 months prior to starting treatment.
5. History of intra-abdominal abscess within 3 months prior to starting treatment (randomisation).
6. History of GI perforation. Patients with a history of abdominal fistula will be considered eligible if the fistula was surgically repaired, there has been no evidence of fistula for at least 6 months prior to starting treatment, and patient is deemed to be at low risk of recurrent fistula.
7. Symptomatic or clinically significant inflammatory bowel disease (Crohn's disease or ulcerative colitis).
8. Patients with an ileostomy will be excluded.
9. Evidence of severe or uncontrolled cardiac disease.

   1. Myocardial infarct or unstable angina within the last 6 months
   2. New York Health Association (NHYA) ≥ grade 2 congestive heart failure
   3. Cardiac ventricular arrhythmias requiring medication
   4. History of 2nd or 3rd degree atrioventricular conduction defects
10. Resting ECG with QTcF > 470msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
11. Evidence of active bleeding or bleeding diathesis.

    Significant haemorrhage of >30ml in a single episode within the last 3 months or any haemoptysis (>5ml fresh blood in last 4 weeks).
12. Malignancy treated within the last 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS) of the breast, Stage 1, grade 1 endometrial carcinoma.
13. Previous treatment with VEGFR tyrosine kinase inhibitors or PARP inhibitors are not permitted.
14. Patients with a known hypersensitivity to excipients of cediranib or olaparib.
15. Persisting ≥ grade 2 CTCAE toxicity (except alopecia and neuropathy) from previous anti-cancer treatment.
16. Major surgery within 14 days before anticipated start of treatment and patients must have recovered from any effects of major surgery.
17. Inability to attend or comply with treatment or follow-up scheduling.
18. Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contra-indicated the use of an investigation drug or puts the patients at high risk for treatment-related complications.
19. Pregnant or breast-feeding women are excluded. Women of childbearing potential will be excluded unless effective methods of contraception are used from signing of the informed consent, throughout the period of taking study treatment and for at least 6 weeks after last dose of trial drug(s).
20. Treatment with any other investigational agent, or participation in another interventional clinical trial within 28 days prior to enrolment (randomisation).
21. Concomitant use of known strong CYP3A4 inhibitors (such as systemic ketoconazole, itraconazole, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir, telithromycin and clarithromycin or moderate CYP3A inhibitors (e.g. systemic Ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
22. Concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
23. Patients with myelodysplastic syndrome/acute myeloid leukaemia.
24. Other psychological, psychiatric, social or medical condition, physical examination finding or a laboratory abnormality that the Investigator considers would make the patient a poor trial candidate or could interfere with protocol compliance or the interpretation of trial results.
25. Patients with known active hepatitis (i.e. Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids.
26. Immunocompromised patients e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV) and are receiving antiviral therapy.
27. Patients with symptomatic uncontrolled brain or meningeal metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment.
28. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
29. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2018-06-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) measured from the date of randomisation to the date of objective progression (investigator assessed using RECIST v1.1) or date of death from any cause (in the absence of progression) | 3 years
  Progression free survival (PFS) measured from the time of randomisation.

SECONDARY OUTCOMES:
Toxicity | 3 years
  Toxicity (AEs) experienced by patients as assessed by the Common Terminology Criteria for Adverse Events v4.03
PFS and OS measured from the time of starting chemotherapy | 3 years
  PFS and OS measured from the time of starting chemotherapy
Adherence to maintenance therapy- compliance and dose reductions and interruptions | 3 years
  Adherence to maintenance therapy- compliance and dose reductions and interruptions
TSST (the time from randomisation to start of second subsequent therapy or death) | 3 years
  TSST (the time from randomisation to start of second subsequent therapy or death)
Quality of life using EORTC QLQ C30 | 3 years
  Quality of life using EORTC QLQ C30
Quality of life using EORTC QLQ OV28 | 3 years
  Quality of life using EORTC QLQ OV28
Cost effectiveness using EQ-5D-5L for economic evaluation | 3 years
  Cost effectiveness using EQ-5D-5L for economic evaluation
VIII. Response rate (RECIST v1.1 and/or CA125) at 16 weeks of treatment in patients who had RECIST v1.1 measurable disease or elevated CA125 at randomisation. RECIST measurements will be based on investigator assessment not central review | 3 years
  VIII. Response rate (RECIST v1.1 and/or CA125) at 16 weeks of treatment in patients who had RECIST v1.1 measurable disease or elevated CA125 at randomisation. RECIST measurements will be based on investigator assessment not central review
Overall survival (OS) measured from the date of randomisation to the date of death from any cause | 3 years
  Overall survival (death from any cause) measured from the time of randomisation.

CONTACTS AND LOCATIONS:
Locations (54):
- Australia (16):
  - Calvary Mater Hospital, Sydney, New South Wales
  - Campbelltown Hospital, Sydney, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Royal Hobart Hospital, Hobart, Tasmania
  - Border Medical Oncology, Albury
  - Flinders Medical Centre, Bedford Park
  - Pindara Private Hospital, Benowa
  - Chris O'Brien Lifehouse, Camperdown
  - Canberra Hospital, Canberra
  - Monash Health, Clayton
  - Gosford Hospital, Gosford
  - Peter MacCallum Cancer Centre, Melbourne
  - ICON Cancer Centre, South Brisbane
  - Mater Cancer Centre, South Brisbane
  - Townsville Hospital, Townsville
  - Westmead Hospital, Westmead
- Canada (7):
  - Cross Cancer Institute, Edmonton
  - Centre Hospitalier de L'Universite de Montreal, Montreal
  - CHU de Quebec, Québec
  - Princess Margaret Cancer Centre, Toronto
  - Sunnybrook Hospital, Toronto
  - BC Cancer Vancouver, Vancouver
  - BC Cancer Victoria, Victoria
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
- United Kingdom (29):
  - Furness General Hospital, Barrow in Furness
  - Belfast City Hospital, Belfast
  - Royal Sussex County Hospital, Brighton
  - Addenbrookes Hospital, Cambridge
  - Kent & Canterbury Hospital, Canterbury
  - Velindre Cancer Centre, Cardiff
  - Cheltenham General Hospital, Cheltenham
  - University Hospital Coventry, Coventry
  - Ninewells Hospital, Dundee
  - Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Surrey County Hospital, Guildford
  - Royal Lancaster Infirmary, Lancaster
  - Guy's Hospital, London
  - Hammersmith Hospital, London
  - Mount Vernon Cancer Centre, London
  - Royal Marsden NHS Foundation Trust, London
  - University College London Hospital, London
  - The Christie Hospital, Manchester
  - Queen Elizabeth the Queen Mother Hospital, Margate
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Churchill Hospital, Oxford
  - Queen Alexandra Hospital, Portsmouth
  - Royal Berkshire Hospital, Reading
  - Southampton General Hospital, Southampton
  - Lister Hospital, Stevenage
  - Singleton Hospital, Swansea
  - Musgrove Park Hospital, Taunton
  - Royal Cornwall, Truro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Elyashiv O, Ledermann J, Parmar G, Farrelly L, Counsell N, Feeney A, El-Khouly F, Macdonald I, Neto A, Arthur-Darkwa E, Burnett E, Jayson GC, Mileshkin L, Gourley C, Nicum S. ICON 9-an international phase III randomized study to evaluate the efficacy of maintenance therapy with olaparib and cediranib or olaparib alone in patients with relapsed platinum-sensitive ovarian cancer following a response to platinum-based chemotherapy. Int J Gynecol Cancer. 2021 Jan;31(1):134-138. doi: 10.1136/ijgc-2020-002073. Epub 2020 Oct 23. PMID 33097567